CLINICAL TRIAL: NCT04199741
Title: Immuno-PET Imaging of Neuroendocrine Tumors Using 89Zr-DFO-SC16.56, a DLL3-targeting Monoclonal Antibody
Brief Title: PET/CT Imaging of Small Cell Lung Cancer Using 89Zr-DFO-SC16.56
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-292
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Small cell lung cancer; Small Cell Lung Carcinoma; 89Zr-DFO-SC16.56; 19-292; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Up to 12 participants with tumors that are found to be >/= 50% positive for DLL3 by IHC
  Interventions: Drug: 89Zr-DFO-SC16.56; Drug: SC16.56, Phase I, Cohort 2; Drug: SC16.56, Phase I, Cohort 3
- Phase II (Experimental): Up to 18 participants with tumors that are found to be >/= 50% positive for DLL3 by IHC
  Interventions: Drug: 89Zr-DFO-SC16.56; Drug: SC16.56, Phase II

INTERVENTIONS:
Drug: 89Zr-DFO-SC16.56 — Injection of 2 mCi of 89Zr-DFO-SC16.56 for Phase I participants. Dose for Phase II will be determined by results from Phase I.
Drug: SC16.56, Phase I, Cohort 2 — 7.5mg
  Arms: Phase I
Drug: SC16.56, Phase I, Cohort 3 — 22.5mg
  Arms: Phase I
Drug: SC16.56, Phase II — Dose for Phase II will be determined by results from Phase I.
  Arms: Phase II

SUMMARY:
The purpose of this study is to look at how safe 89Zr-DFO-SC16.56 is, and how it is processed by the body in people with small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent
* Age 4 or more years
* Histologically confirmed, SCLC, (newly diagnosed or recurrent); small cell carcinoma of unknown or non-lung origin; or other types of neuroendocrine tumor OR
* Histologically confirmed prostate cancer, with suspected or confirmed NEPC based upon clinical assays obtained prior to the trial OR
* Histologically confirmed or suspected primary brain neoplasm
* Desmoplastic small round cell tumors, osteosarcoma, Ewing's sarcoma, rabdomyosarcoma, Wilms tumors, hepatoblastomas, rhabdoid tumors and neuroblastoma patients
* At least one tumor lesion on CT2 or MRI ≥ 0.8 cm OR
* Tumor detectable FDG PET, PSMA PET, DOTATATE PET, MIBG SPECT (or planar MIBG scan if SPECT unavailable) OR
* MRI or bone scan that shows new osseous metastases. The scans should have been obtained in the last 12 weeks
* ECOG performance status 0 to 2
* Performance Status: Subjects must have a Lansky (<16 years of at least 40)
* Negative serum pregnancy test within 2 weeks of 89Zr- DFO-SC16.56 or women of child-bearing potential

  * Available archival tumor specimen suitable for DLL3 IHC or clinician already has plans to obtain tumor specimen as part of standard of care (unrelated to patient participation in 19-292) which will yield sufficient tumor specimen to allow for DLL3 IHC
  * For the prostate cancer patient cohort with only bone metastases, a recent PET scan (FDG or PSMA-targeted) that shows tracer-avid osseous metastases, a recent MRI that shows new osseous metastases, a bone scan that shows new osseous metastases, or have recent PET or SPECT scans that demonstrate tumors that are evaluable by PET or SPECT. The scans should have been obtained in the last 8 weeks.

    1. Patients with SCLC will be the primary study population, however patients with other types of neuroendocrine tumors may be included at the PI's discretion.
    2. Criterion is intended to demonstrate presence of imageable disease. A low-dose CT (e.g. from a PET/CT scan) may be used at PI's discretion.
    3. While willingness to undergo the biopsy is required if archival tissue is not available, PET/CT guided biopsy is not a mandatory study assessment. As described in section 9.3, the guided biopsy may be waived at the discretion of the principal investigator if the DLL3 PET/CT reveals no sites of DLL3 tracer-avid tumor or if the principal investigator deems it is not in the best interest of the patient, according to best clinical judgement. The pediatric population would not be approached for an optional PET/CT-guided biopsy

Exclusion Criteria:

* History of anaphylactic reaction to humanize or human antibodies
* Pregnant or breast feeding
* Psychiatric illness that would interfere with compliance with the study procedures
* Inability to undergo PET scan due to weight limit
* Patients who require anesthesia or monitored sedation to tolerate PET scan procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Phase I: Radiation Dosimetry of 89Zr- DFO-SC16.56 PET/CT imaging in participants | Up to 12 months
  The PET and blood data are used to quantify tracer-biodistribution, measuring the amount of radioactivity present in the blood and bodily regions-of-interest
Phase I: Safety of 89Zr- DFO-SC16.56 PET/CT imaging in cancer patients by evaluating toxicities | up to 12 months
  89Zr- DFO-SC16.56 PET/CT will be considered safe if there are no possibly probably, or definitely related grade 3 or higher toxicities (except allergic reactions) among the patients enrolled in the phase I portion
Phase II: Correlation between tumor uptake of 89Zr- DFO-SC16.56 with expression of DLL3 | Up to 12 months
  This is determined by immunohistochemistry and quantitative mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Dunphy, DO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Tendler S, Dunphy MP, Agee M, O'Donoghue J, Aly RG, Choudhury NJ, Kesner A, Kirov A, Mauguen A, Baine MK, Schoder H, Weber WA, Rekhtman N, Lyashchenko SK, Bodei L, Morris MJ, Lewis JS, Rudin CM, Poirier JT. Imaging with [89Zr]Zr-DFO-SC16.56 anti-DLL3 antibody in patients with high-grade neuroendocrine tumours of the lung and prostate: a phase 1/2, first-in-human trial. Lancet Oncol. 2024 Aug;25(8):1015-1024. doi: 10.1016/S1470-2045(24)00249-3. Epub 2024 Jun 28. PMID 38950555
- [Derived] Tully KM, Tendler S, Carter LM, Sharma SK, Samuels ZV, Mandleywala K, Korsen JA, Delos Reyes AM, Piersigilli A, Travis WD, Sen T, Pillarsetty N, Poirier JT, Rudin CM, Lewis JS. Radioimmunotherapy Targeting Delta-like Ligand 3 in Small Cell Lung Cancer Exhibits Antitumor Efficacy with Low Toxicity. Clin Cancer Res. 2022 Apr 1;28(7):1391-1401. doi: 10.1158/1078-0432.CCR-21-1533. PMID 35046060
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org